CLINICAL TRIAL: NCT02317523
Title: Alzheimer's Caregiver Coping: Mental and Physical Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Brent Mausbach, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMausbach; RF1AG015301 (NIH)
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease; Alzheimer Dementia; Alzheimer's Disease; Dementia
Keywords: Dementia; Caregiver; Cardiovascular Disease; Stress; Depression; Anxiety; Heart Disease; Carer; Care Giver; Caregiving; Psychotherapy; Therapy; Behavioral Activation; Education; Intervention; CBT; Cognitive-Behavior Therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cardiovascular Diseases; Depression; Anxiety Disorders; Heart Diseases | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Activation (Experimental): Behavioral Activation (BA) emphasize self-monitoring as an aid for increasing one's engagement in self-reinforcing activities while simultaneously reducing negative avoidant coping responses. The intervention consists of 6 total face-to-face sessions lasting 60 minutes each.
  Interventions: Behavioral: Behavioral Activation
- Information and Support (Active Comparator): Information and Support (IS) consists of providing education on Alzheimer's disease, coping with specific stresses prevalent in caregiving, and community-based services available for caregivers. Caregivers choose information most relevant to their current circumstances, and can discuss this with their counselor during the sessions. In addition, the IS condition encompasses elements of supportive therapy including empathy and active listening. The intervention consists of 6 total face-to-face sessions lasting 60 minutes each.
  Interventions: Behavioral: Information and Support

INTERVENTIONS:
Behavioral: Behavioral Activation — Six face-to-face sessions (60 minutes each) of Behavioral Activation (BA) therapy
  Arms: Behavioral Activation
Behavioral: Information and Support — Six face-to-face sessions (60 minutes each) of Supportive Therapy
  Arms: Information and Support

SUMMARY:
This study evaluates the effectiveness of Behavioral Activation (BA) therapy vs Support and Information for reducing risk for emotional and cardiovascular diseases in Alzheimer's caregivers. Half of participants will receive BA and the other half will receive support and information.

DETAILED DESCRIPTION:
The burden of caring for a loved-one with Alzheimer's disease is associated with adverse psychological and general health consequences for the caregiver. These consequences including risk for depression, cardiovascular disease, and earlier mortality. Because preliminary work has demonstrated that an educational programs for caregivers reduce the negative affect associated with caregiving, the investigators wish to determine whether improving mood can also modify pathophysiological changes that have been linked to risk for developing cardiovascular disease.

The investigators aims are to determine whether a 6-week Behavioral Activation (BA) intervention, followed by 3 booster sessions over a period of 6 months, compared to an Information-Support (IS) intervention will be associated with significant improvement in indicators of vascular pathology, modification of psychobiological markers that have been associated with cardiovascular parameters, and to determine whether improvements in indicators of vascular parameters will be mediated by treatment related change in measures of distress and markers of cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or older.
* Providing in-home care to a spouse with dementia.

Exclusion Criteria:

* Taking Coumarin anticoagulants.
* Taking nitrates or niacin.
* Taking non-selective β-blockers.
* Glucocorticoid use in the 2 weeks prior to enrollment.
* Taking Aldomet or labetalol.
* Neither the caregiver nor Alzheimer's patient can be diagnosed with a terminal illness with a life expectancy of less than 1 year
* Cognitive impairment
* Caregivers enrolled in another intervention study or receiving psychotherapy to improve well-being or reduce distress
* Blood pressure >200/120 mm Hg

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-09; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent Flow Mediated Dilation (FMD) | Change from baseline to 2-year follow-up
  Flow-Mediated Dilation
Center for Epidemiologic Studies - Depression (CES-D) scale | Change from baseline to 2-year follow-up
  Depressive Symptoms
Interleukin-6 | Change from baseline to 2-year follow-up
  Inflammation (IL-6)

SECONDARY OUTCOMES:
Baroreflex Sensitivity (BRS) | Change from baseline to 2-year follow-up
  Arterial function (baroreceptors)
Arterial Compliance (AC) | Change from baseline to 2-year follow-up
  Arterial function
Carotid Intima Media Thickness (IMT) | Change from baseline to 2-year follow-up
  Vascular outcome
D-dimer | Change from baseline to 2-year follow-up
  Coagulation
C-reactive Protein (CRP) | Change from baseline to 2-year follow-up
  Inflammation
Tumor Necrosis Factor (TNF)- alpha | Change from baseline to 2-year follow-up
  Biomarker
Plasminogen Activator Inhibitor (PAI)-1 | Change from baseline to 2-year follow-up
  Coagulation
von Willebrand Factor (vWF) | Change from baseline to 2-year follow-up
  Coagulation

CONTACTS AND LOCATIONS:
Overall Officials: Brent T Mausbach, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] von Kanel R, Mausbach BT, Dimsdale JE, Ziegler MG, Mills PJ, Allison MA, Patterson TL, Ancoli-Israel S, Grant I. Refining caregiver vulnerability for clinical practice: determinants of self-rated health in spousal dementia caregivers. BMC Geriatr. 2019 Jan 22;19(1):18. doi: 10.1186/s12877-019-1033-2. PMID 30669980